CLINICAL TRIAL: NCT00115492
Title: A Randomized, Double-Blind, Parallel Group, 52-Week Study to Compare the Effect of Fluticasone Propionate/Salmeterol Diskus Combination Product 250/50mcg BID With Salmeterol Diskus 50mcg BID on the Annual Rate of Moderate/Severe Exacerbations in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Advair® DISKUS® Versus Serevent® DISKUS® For Chronic Obstructive Pulmonary Disease Exacerbations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO100250
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Breathing; Exacerbation; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluticasone Propionate/Salmeterol Combination Product
Drug: Salmeterol
  Other Names: Fluticasone Propionate/Salmeterol Combination Product

SUMMARY:
This study evaluates the effect of two medicines on COPD (Chronic Obstructive Pulmonary Disease) exacerbations. This study will last up to 56 weeks, and subjects will visit the clinic 10 times. Subjects will be given breathing tests and will record their breathing symptoms daily on diary cards. All study related medicines and medical examinations will be provided at no cost. The two drugs used in this study have been approved by FDA for use in patients with COPD.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel Group, 52-week Study to Compare the Effect of the Fluticasone Propionate/Salmeterol DISKUS Combination Product 250/50mcg BID with Salmeterol DISKUS 50mcg BID on the Annual Rate of Moderate/Severe Exacerbations in Subjects with Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD.
* Current or previous cigarette smokers with a smoking history of at least 10 pack-years.
* History of at least 1 COPD exacerbation in the 12 months prior to screening.
* Forced expiratory volume in one second (FEV1) of less than or equal to 50% of predicted normal.

Exclusion criteria:

* Diagnosis of asthma.
* Additional respiratory disorders other than COPD (eg, sarcoidosis, alpha-1 antitrypsin deficiency, cystic fibrosis, or active tuberculosis).
* Concurrent use of long-acting beta-agonists, long-acting anticholinergics, inhaled and oral corticosteroids, theophylline, investigational medications, ritonavir, and anti-leukotrienes.
* Lung resection surgery within 1 year of screening.
* Abnormal and clinically significant ECG findings at screening.
* Other inclusion and exclusion criteria will be evaluated at the first study visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2004-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Rate of moderate/severe exacerbations over a 52 week treatment period

SECONDARY OUTCOMES:
The time until the first moderate/severe exacerbation; the annual rate of exacerbations requiring oral corticosteroid treatment, and breathing tests conducted over one year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (91):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Olathe, Kansas
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Absecon, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Bay Shore, New York
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Larchmont, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Chardon, Ohio
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, McKeesport, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (15):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Holyrood, Newfoundland and Labrador
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Charlesbourg, Quebec
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Saint-Léonard, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Disantostefano RL, Li H, Rubin DB, Stempel DA. Which patients with chronic obstructive pulmonary disease benefit from the addition of an inhaled corticosteroid to their bronchodilator? A cluster analysis. BMJ Open. 2013 Apr 22;3(4):e001838. doi: 10.1136/bmjopen-2012-001838. Print 2013. PMID 23613569
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO100250 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register